CLINICAL TRIAL: NCT06841185
Title: A Randomized, Multicenter, Double-Blind, Parallel-Controlled Integrated Phase I/III Clinical Study to Evaluate the Efficacy, Safety, Immunogenicity, and Pharmacokinetic Profile of Ipilimumab Biosimilar HLX13 Vs. YERVOY® (US-Sourced YERVOY® and EU-Sourced YERVOY®) As a First-Line Treatment for Patients with Unresectable Hepatocellular Carcinoma
Brief Title: A Study to Compare the Efficacy, Safety, Immunogenicity, and Pharmacokinetic Profile of HLX13 with YERVOY As a First-Line Treatment for Patients with Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX13-HCC301
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Ipilimumab Biosimilar
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HLX13 group (Experimental): Recombinant anti-CTLA-4 fully human monoclonal antibody injection developed by Shanghai Henlius Biotech, Inc.
  Interventions: Drug: HLX13
- US-sourced YERVOY® group (Active Comparator): US-sourced ipilimumab
  Interventions: Drug: US-sourced YERVOY®
- EU-sourced YERVOY® group (Active Comparator): EU-sourced ipilimumab
  Interventions: Drug: EU-sourced YERVOY®

INTERVENTIONS:
Drug: HLX13 — HLX13 (3 mg/kg) and nivolumab (1 mg/kg) treatment on the first day of each cycle, every 3 weeks with a total of 4 cycles
  Arms: HLX13 group
Drug: US-sourced YERVOY® — US-sourced YERVOY® (3 mg/kg) and nivolumab (1 mg/kg) treatment on the first day of each cycle, every 3 weeks with a total of 4 cycles
  Arms: US-sourced YERVOY® group
Drug: EU-sourced YERVOY® — EU-sourced YERVOY® (3 mg/kg) and nivolumab (1 mg/kg) treatment on the first day of each cycle, every 3 weeks with a total of 4 cycles
  Arms: EU-sourced YERVOY® group

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-controlled integrated phase I/III clinical study to evaluate the efficacy, safety, PK, and immunogenicity of HLX13 and YERVOY® in patients with unresectable hepatocellular carcinoma who have not received prior systemic therapy.

DETAILED DESCRIPTION:
This study includes three treatment groups. Patients will be randomly assigned at a 2:1:1 ratio to the HLX13, US-sourced YERVOY®, or EU-sourced YERVOY® group to receive the treatment of IMPs in combination with nivolumab.

Patients with good tolerability and disease control will receive HLX13 or YERVOY® in combination with nivolumab on the first day of every 3 weeks for up to 4 cycles. PK and immunogenicity blood sampling will be conducted during the treatment period. After the four treatment cycles, all subjects will be subsequently treated with nivolumab monotherapy until investigator-assessed disease progression, initiation of a new anti-neoplastic therapy, withdrawal of informed consent, death, unacceptable toxicity, or up to 1 year after randomization, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed relapsed metastatic or advanced hepatocellular carcinoma not eligible for surgical or locoregional therapies according to the diagnostic criteria of the American Association for the Study of Liver Diseases (AASLD).
* At least one measurable lesion as assessed by IRRC based on RECIST v1.1 within 4 weeks prior to the first dose in this study.
* No systemic therapy for relapsed metastatic or advanced hepatocellular carcinoma prior to screening.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Child-Pugh Class A.
* Normal major organ functions.
* Women of childbearing potential should use highly effective methods of contraception during the study and within 5 months after the last study treatment; Male subjects capable of fathering a child must agree to use at least one highly effective method of contraception for the duration of the study and for at least 7 months after the last study treatment.

Exclusion Criteria:

* With other histopathological types of hepatocellular carcinoma.
* History of hepatic encephalopathy.
* Clinically significant ascites.
* Patients with tumor thrombus at the main portal vein, left or right portal (either or both) vein branch, or inferior vena cava.
* Presence of the central nervous system disorders at screening, except subjects who have previously received treatment for brain metastases can participate in the study treatment if their clinical symptoms have been stable for at least 4 weeks.
* Evidence of portal hypertension with bleeding esophageal or gastric varices within 6 months prior to the randomization.
* Known active or suspected autoimmune diseases.
* Active co-infection with both hepatitis B and C, or hepatitis D infection in subjects with hepatitis B.
* Uncontrolled cardiovascular diseases within 6 months.
* Known interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, and severe lung function abnormalities that may impede the investigators' diagnosis and management of drug-related pulmonary toxicity prior to screening.
* Patients who have received any T-cell costimulatory agents or immune checkpoint blockade therapy, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other agents that target T cells.
* Patients who have other conditions not suitable for inclusion per investigator's judgments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-06-06 (Estimated); Study Completion 2028-05-05 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to 21 days (AUC0-21d) | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Area under the serum concentration-time curve within a dosing interval at steady-state (AUCss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Best Objective Response Rate (ORR) up to Week 24 (assessed by Independent Radiology Review Committee [IRRC] based on RECIST v1.1) | Up to Week 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Maximum serum drug concentration (Cmax) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Trough serum drug concentration (Ctrough) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum serum drug concentration (Tmax) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Elimination half-life (t1/2) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Total clearance (CL) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Volume of distribution during terminal phase (Vz) after the first dose | Up to Day 21
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum serum drug concentration at steady state (Tmax, ss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Maximum serum drug concentration at steady state (Cmax, ss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Minimum serum drug concentration at steady state (Cmin, ss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Elimination half-life (t1/2) at steady state | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Volume of distribution at steady state (Vss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Total clearance at steady state (CLss) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Accumulation ratio of AUC (Rac, AUC) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Accumulation ratio of Cmax (Rac, Cmax) | Up to Day 85
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
ORR assessed by IRRC (based on RECIST v1.1) | Up to Week 30
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
ORR assessed by investigators (based on RECIST v1.1) | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Duration of Response (DOR) assessed by investigators (based on RECIST v1.1) | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to Response (TTR) assessed by investigators (based on RECIST v1.1) | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Progression-Free Survival (PFS) Status assessed by investigators (based on RECIST v1.1) | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Progression-Free Survival Rate (PFSR) assessed by investigators (based on RECIST v1.1) at Weeks 24 and 48 | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Overall Survival (OS) | Up to 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Overall Survival Rate (OSR) assessed by investigators (based on RECIST v1.1) at Weeks 24 and 48 | Up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Adverse events (AEs) | Up to Month 15
Serious adverse events (SAEs) | Up to Month 15
Incidence of anti-drug antibodies (ADAs). | Up to 1 year
Incidence of neutralizing antibodies (NAbs). | Up to 1 year

IPD SHARING:
Plan to Share IPD: No